CLINICAL TRIAL: NCT00691080
Title: Characterization of Endogenous Melatonin Profiles in Children With Autism Spectrum Disorder.
Brief Title: Understanding Sleep Problems in Children With Autism Spectrum Disorder
Acronym: REST
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Autism Speaks (Other); Oregon Health and Science University (Other); Columbia University (Other); The Emmes Company, LLC (Industry); Autism Treatment Network (Network)
Responsible Party: Principal Investigator, Daniel Glaze, Principal Investigator, Baylor College of Medicine
Other Study IDs: 2003
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Sleep Problems
Keywords: Melatonin; Sleep; Autism; ASD; Sleep problems in children with autism spectrum disorder
MeSH Terms: conditions — Parasomnias; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — SAMPLE: Saliva What is the purpose of the sample collection? Determination of dim light melatonin onset (DMLO), as measured by salivary melatonin secretion.
  SAMPLE: Urine What is the purpose of the sample collection? Measurement of secreted 6-suplhatoxymaltonin, a metabolite of melatonin.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ASD children: ASD children as defined by:
  1. Age greater than or equal to 4 or less than or equal to 9 years
  2. Diagnosis of Autism Spectrum Disorder; supported by ADOS and the ADI or SCQ (subjects).
  3. No current use of psychoactive medications (e.g. fluoxetine, methylphenidate, risperidone, lithium, etc.)
  4. No current or use within the last 1 month of beta-blockers or melatonin
  5. No current use of sleep aids
  6. No presence of untreated medical problems that could otherwise explain sleep problems (e.g. obstructive sleep apnea, gastroesophageal reflux disease - GERD)
  (6) No blindness.
- "Healthy" control children: "Healthy" control children as defined by:
  1. Age greater than or equal to 4 or less than or equal to 9 years
  2. A SCQ score of less than 10 without parental or physician concern for another neurodevelopmental disorder will be used to define normal children.
  3. No current use of psychoactive medications (e.g. fluoxetine, methylphenidate, risperidone, lithium, etc.)
  4. No current or use within the last 1 month of beta-blockers or melatonin
  5. No current use of sleep aids;
  6. No presence of untreated medical problems that could otherwise explain sleep problems (e.g. obstructive sleep apnea, gastroesophageal reflux disease - GERD)
  (6) No blindness. (7) No current or past diagnosis of ADHD, depression, anxiety or with any other psychiatric conditions.
  (8) No sibling with a diagnosis of Autism Spectrum Disorder.

SUMMARY:
The investigators will examine whether sleep problems in children with autism spectrum disorder (ASD) are related to alterations in the production of melatonin (MT), a hormone that plays an important role in regulating sleep-wake cycle. Children with ASD experience high rates of sleep disturbances that potentially contribute to problems with thinking and behavior. It is unclear if changes in MT production cause sleep problems in children with ASD. MT is frequently used to treat these sleep problems; however, it has not been well established whether MT is an effective treatment. Our hypotheses concerning MT is children with ASD and sleep problems will have a delayed sleep-wake cycle and/or decreased MT production. This study will compare children diagnosed with ASD to "healthy" control children with no ASD diagnosis. All subjects will be recruited from one of three sites: Baylor College of Medicine, Oregon Health & Science University and Columbia University. The investigators will use a standardized questionnaire to determine whether the child has sleep problems. The investigators will measure MT levels in saliva in ASD children with sleep problems and in a group of control children without sleep problems. Total 24-hour MT production will be determined from urine samples in these same two groups.

DETAILED DESCRIPTION:
This is a proposal to study the relationship between melatonin (MT) and sleep problems in children with autism spectrum disorder (ASD), as part of the collaborative research structure of the Autism Treatment Network (ATN). A major goal of the ATN is to conduct clinical research that will have a significant impact on the daily lives and functioning of individuals with ASD and to address immediate concerns of parents. Children with ASD experience high rates of sleep disturbance, which likely contribute to the severity of their daytime cognitive and behavioral dysfunction and to poorer quality of life for them and their families.

As a step toward addressing sleep problems in ASD, we propose to test the hypothesis that children with ASD and sleep problems will have a delay in MT onset and/or have decreased MT secretion over 24 hours compared to normal controls.

Primary endpoint: Characterize the endogenous MT profiles in children with ASD:

We predict that results from this study will reveal lower levels of metabolized MT in children with ASD when compared to normal children. In addition, we anticipate that children with ASD will have delayed MT onset or altered circadian phase.

Data from this study will provide important information concerning circadian rhythm dysregulation in ASD and will support the development of future studies using MT to modify and correct abnormal circadian rhythms.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Autism Spectrum Disorder; supported by ADOS and the ADI or SCQ (subjects).
2. Age greater than or equal to 4 or less than or equal to 9 years;
3. Parents have given informed consent.
4. Parent/Caregiver fluent in written and spoken English.
5. Controls only: A SCQ score of less than 10 without parental or physician concern for another neurodevelopmental disorder will be used to define normal children.

Exclusion Criteria:

1. Current use of psychoactive medications (e.g. fluoxetine, methylphenidate, risperidone, lithium, etc.)*;
2. Current or use within the last 1 month of beta-blockers or melatonin;
3. Current use of sleep aids;
4. Presence of untreated medical problems that could otherwise explain sleep problems (e.g. obstructive sleep apnea, gastroesophageal reflux disease - GERD);
5. Blindness.
6. Controls only: current or past diagnosis of ADHD, depression, anxiety or with any other psychiatric conditions. (7) Controls only: Sibling has a diagnosis of Autism Spectrum Disorder.

   * Psychoactive medications can be discontinued but the parents must discuss medication discontinuation with their prescribing physician prior to reducing or stopping the medications.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with the diagnosis of ASD and that are not diagnosised with ASD (controls).
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Sleep Latency, as measured by actigraphy | 1 week

SECONDARY OUTCOMES:
Total sleep time, as measured by actigraphy | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Glaze, M.D., Study Director — Baylor College of Medicine
Locations (3):
- United States (3):
  - Columbia University, New York, New York
  - Oregon Health & Sciences University, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Couturier JL, Speechley KN, Steele M, Norman R, Stringer B, Nicolson R. Parental perception of sleep problems in children of normal intelligence with pervasive developmental disorders: prevalence, severity, and pattern. J Am Acad Child Adolesc Psychiatry. 2005 Aug;44(8):815-22. doi: 10.1097/01.chi.0000166377.22651.87. PMID 16034284
- [Background] Wiggs L, Stores G. Severe sleep disturbance and daytime challenging behaviour in children with severe learning disabilities. J Intellect Disabil Res. 1996 Dec;40 ( Pt 6):518-28. doi: 10.1046/j.1365-2788.1996.799799.x. PMID 9004112
- [Background] Patzold LM, Richdale AL, Tonge BJ. An investigation into sleep characteristics of children with autism and Asperger's Disorder. J Paediatr Child Health. 1998 Dec;34(6):528-33. doi: 10.1046/j.1440-1754.1998.00291.x. PMID 9928644
- [Background] Richdale AL, Prior MR. The sleep/wake rhythm in children with autism. Eur Child Adolesc Psychiatry. 1995 Jul;4(3):175-86. doi: 10.1007/BF01980456. PMID 8846206
- [Background] Fallone G, Acebo C, Arnedt JT, Seifer R, Carskadon MA. Effects of acute sleep restriction on behavior, sustained attention, and response inhibition in children. Percept Mot Skills. 2001 Aug;93(1):213-29. doi: 10.2466/pms.2001.93.1.213. PMID 11693688
- [Background] Polimeni MA, Richdale AL, Francis AJ. A survey of sleep problems in autism, Asperger's disorder and typically developing children. J Intellect Disabil Res. 2005 Apr;49(Pt 4):260-8. doi: 10.1111/j.1365-2788.2005.00642.x. PMID 15816813
- [Background] Giannotti F, Cortesi F, Cerquiglini A, Bernabei P. An open-label study of controlled-release melatonin in treatment of sleep disorders in children with autism. J Autism Dev Disord. 2006 Aug;36(6):741-52. doi: 10.1007/s10803-006-0116-z. PMID 16897403
- [Background] Allik H, Larsson JO, Smedje H. Insomnia in school-age children with Asperger syndrome or high-functioning autism. BMC Psychiatry. 2006 Apr 28;6:18. doi: 10.1186/1471-244X-6-18. PMID 16646974
- [Background] Hoshino Y, Watanabe H, Yashima Y, Kaneko M, Kumashiro H. An investigation on sleep disturbance of autistic children. Folia Psychiatr Neurol Jpn. 1984;38(1):45-51. doi: 10.1111/j.1440-1819.1984.tb00353.x. PMID 6537391
- [Background] Clements J, Wing L, Dunn G. Sleep problems in handicapped children: a preliminary study. J Child Psychol Psychiatry. 1986 May;27(3):399-407. doi: 10.1111/j.1469-7610.1986.tb01841.x. PMID 3733919
- [Background] Quine L. Sleep problems in children with mental handicap. J Ment Defic Res. 1991 Aug;35 ( Pt 4):269-90. doi: 10.1111/j.1365-2788.1991.tb00402.x. PMID 1757978
- [Background] Honomichl RD, Goodlin-Jones BL, Burnham M, Gaylor E, Anders TF. Sleep patterns of children with pervasive developmental disorders. J Autism Dev Disord. 2002 Dec;32(6):553-61. doi: 10.1023/a:1021254914276. PMID 12553592
- [Background] Schreck KA, Mulick JA. Parental report of sleep problems in children with autism. J Autism Dev Disord. 2000 Apr;30(2):127-35. doi: 10.1023/a:1005407622050. PMID 10832777
- [Background] Wiggs L, Stores G. Sleep patterns and sleep disorders in children with autistic spectrum disorders: insights using parent report and actigraphy. Dev Med Child Neurol. 2004 Jun;46(6):372-80. doi: 10.1017/s0012162204000611. PMID 15174528
- [Background] Didden R, Korzilius H, van Aperlo B, van Overloop C, de Vries M. Sleep problems and daytime problem behaviours in children with intellectual disability. J Intellect Disabil Res. 2002 Oct;46(Pt 7):537-47. doi: 10.1046/j.1365-2788.2002.00404.x. PMID 12354310
- [Background] Robinson AM, Richdale AL. Sleep problems in children with an intellectual disability: parental perceptions of sleep problems, and views of treatment effectiveness. Child Care Health Dev. 2004 Mar;30(2):139-50. doi: 10.1111/j.1365-2214.2004.00395.x. PMID 14961866
- [Background] Bradley EA, Summers JA, Wood HL, Bryson SE. Comparing rates of psychiatric and behavior disorders in adolescents and young adults with severe intellectual disability with and without autism. J Autism Dev Disord. 2004 Apr;34(2):151-61. doi: 10.1023/b:jadd.0000022606.97580.19. PMID 15162934
- [Background] Mindell JA, Emslie G, Blumer J, Genel M, Glaze D, Ivanenko A, Johnson K, Rosen C, Steinberg F, Roth T, Banas B. Pharmacologic management of insomnia in children and adolescents: consensus statement. Pediatrics. 2006 Jun;117(6):e1223-32. doi: 10.1542/peds.2005-1693. PMID 16740821
- [Background] Dahl RE. The impact of inadequate sleep on children's daytime cognitive function. Semin Pediatr Neurol. 1996 Mar;3(1):44-50. doi: 10.1016/s1071-9091(96)80028-3. PMID 8795841
- [Background] Beebe DW, Wells CT, Jeffries J, Chini B, Kalra M, Amin R. Neuropsychological effects of pediatric obstructive sleep apnea. J Int Neuropsychol Soc. 2004 Nov;10(7):962-75. doi: 10.1017/s135561770410708x. PMID 15803560
- [Background] O'Brien LM, Gozal D. Neurocognitive dysfunction and sleep in children: from human to rodent. Pediatr Clin North Am. 2004 Feb;51(1):187-202. doi: 10.1016/s0031-3955(03)00184-6. PMID 15008589
- [Background] Owens JA, Spirito A, McGuinn M, Nobile C. Sleep habits and sleep disturbance in elementary school-aged children. J Dev Behav Pediatr. 2000 Feb;21(1):27-36. doi: 10.1097/00004703-200002000-00005. PMID 10706346
- [Background] Friedman BC, Hendeles-Amitai A, Kozminsky E, Leiberman A, Friger M, Tarasiuk A, Tal A. Adenotonsillectomy improves neurocognitive function in children with obstructive sleep apnea syndrome. Sleep. 2003 Dec 15;26(8):999-1005. doi: 10.1093/sleep/26.8.999. PMID 14746381
- [Background] Kennedy JD, Blunden S, Hirte C, Parsons DW, Martin AJ, Crowe E, Williams D, Pamula Y, Lushington K. Reduced neurocognition in children who snore. Pediatr Pulmonol. 2004 Apr;37(4):330-7. doi: 10.1002/ppul.10453. PMID 15022130
- [Background] Chervin RD, Ruzicka DL, Giordani BJ, Weatherly RA, Dillon JE, Hodges EK, Marcus CL, Guire KE. Sleep-disordered breathing, behavior, and cognition in children before and after adenotonsillectomy. Pediatrics. 2006 Apr;117(4):e769-78. doi: 10.1542/peds.2005-1837. PMID 16585288
- [Background] Nir I, Meir D, Zilber N, Knobler H, Hadjez J, Lerner Y. Brief report: circadian melatonin, thyroid-stimulating hormone, prolactin, and cortisol levels in serum of young adults with autism. J Autism Dev Disord. 1995 Dec;25(6):641-54. doi: 10.1007/BF02178193. PMID 8720032
- [Background] Kulman G, Lissoni P, Rovelli F, Roselli MG, Brivio F, Sequeri P. Evidence of pineal endocrine hypofunction in autistic children. Neuro Endocrinol Lett. 2000;21(1):31-34. PMID 11455326
- [Background] Leibenluft E, Feldman-Naim S, Turner EH, Schwartz PJ, Wehr TA. Salivary and plasma measures of dim light melatonin onset (DLMO) in patients with rapid cycling bipolar disorder. Biol Psychiatry. 1996 Oct 15;40(8):731-5. doi: 10.1016/0006-3223(95)00488-2. PMID 8894065
- [Background] Lewy AJ, Bauer VK, Hasler BP, Kendall AR, Pires ML, Sack RL. Capturing the circadian rhythms of free-running blind people with 0.5 mg melatonin. Brain Res. 2001 Nov 9;918(1-2):96-100. doi: 10.1016/s0006-8993(01)02964-x. PMID 11684046
- [Background] Lewy AJ, Cutler NL, Sack RL. The endogenous melatonin profile as a marker for circadian phase position. J Biol Rhythms. 1999 Jun;14(3):227-36. doi: 10.1177/074873099129000641. PMID 10452335
- [Background] Lewy AJ, Emens J, Sack RL, Hasler BP, Bernert RA. Zeitgeber hierarchy in humans: resetting the circadian phase positions of blind people using melatonin. Chronobiol Int. 2003 Sep;20(5):837-52. doi: 10.1081/cbi-120024215. PMID 14535357
- [Background] Lewy AJ, Emens JS, Sack RL, Hasler BP, Bernert RA. Low, but not high, doses of melatonin entrained a free-running blind person with a long circadian period. Chronobiol Int. 2002 May;19(3):649-58. doi: 10.1081/cbi-120004546. PMID 12069043
- [Background] Voultsios A, Kennaway DJ, Dawson D. Salivary melatonin as a circadian phase marker: validation and comparison to plasma melatonin. J Biol Rhythms. 1997 Oct;12(5):457-66. doi: 10.1177/074873049701200507. PMID 9376644
- [Background] Tordjman S, Anderson GM, Pichard N, Charbuy H, Touitou Y. Nocturnal excretion of 6-sulphatoxymelatonin in children and adolescents with autistic disorder. Biol Psychiatry. 2005 Jan 15;57(2):134-8. doi: 10.1016/j.biopsych.2004.11.003. PMID 15652871
- [Background] Garstang J, Wallis M. Randomized controlled trial of melatonin for children with autistic spectrum disorders and sleep problems. Child Care Health Dev. 2006 Sep;32(5):585-9. doi: 10.1111/j.1365-2214.2006.00616.x. PMID 16919138
- [Background] Weiss MD, Wasdell MB, Bomben MM, Rea KJ, Freeman RD. Sleep hygiene and melatonin treatment for children and adolescents with ADHD and initial insomnia. J Am Acad Child Adolesc Psychiatry. 2006 May;45(5):512-519. PMID 16670647
- [Background] Paavonen EJ, Nieminen-von Wendt T, Vanhala R, Aronen ET, von Wendt L. Effectiveness of melatonin in the treatment of sleep disturbances in children with Asperger disorder. J Child Adolesc Psychopharmacol. 2003 Spring;13(1):83-95. doi: 10.1089/104454603321666225. PMID 12804129
- [Background] Buscemi N, Vandermeer B, Hooton N, Pandya R, Tjosvold L, Hartling L, Baker G, Klassen TP, Vohra S. The efficacy and safety of exogenous melatonin for primary sleep disorders. A meta-analysis. J Gen Intern Med. 2005 Dec;20(12):1151-8. doi: 10.1111/j.1525-1497.2005.0243.x. PMID 16423108
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] Bloom BJ, Owens JA, McGuinn M, Nobile C, Schaeffer L, Alario AJ. Sleep and its relationship to pain, dysfunction, and disease activity in juvenile rheumatoid arthritis. J Rheumatol. 2002 Jan;29(1):169-73. PMID 11824956
- [Background] Aman MG, Singh NN, Stewart AW, Field CJ. The aberrant behavior checklist: a behavior rating scale for the assessment of treatment effects. Am J Ment Defic. 1985 Mar;89(5):485-91. PMID 3993694
- [Background] McCracken JT, McGough J, Shah B, Cronin P, Hong D, Aman MG, Arnold LE, Lindsay R, Nash P, Hollway J, McDougle CJ, Posey D, Swiezy N, Kohn A, Scahill L, Martin A, Koenig K, Volkmar F, Carroll D, Lancor A, Tierney E, Ghuman J, Gonzalez NM, Grados M, Vitiello B, Ritz L, Davies M, Robinson J, McMahon D; Research Units on Pediatric Psychopharmacology Autism Network. Risperidone in children with autism and serious behavioral problems. N Engl J Med. 2002 Aug 1;347(5):314-21. doi: 10.1056/NEJMoa013171. PMID 12151468
- [Background] Amminger GP, Berger GE, Schafer MR, Klier C, Friedrich MH, Feucht M. Omega-3 fatty acids supplementation in children with autism: a double-blind randomized, placebo-controlled pilot study. Biol Psychiatry. 2007 Feb 15;61(4):551-3. doi: 10.1016/j.biopsych.2006.05.007. Epub 2006 Aug 22. PMID 16920077
- [Background] Shea S, Turgay A, Carroll A, Schulz M, Orlik H, Smith I, Dunbar F. Risperidone in the treatment of disruptive behavioral symptoms in children with autistic and other pervasive developmental disorders. Pediatrics. 2004 Nov;114(5):e634-41. doi: 10.1542/peds.2003-0264-F. Epub 2004 Oct 18. PMID 15492353
- [Background] Scahill L, Aman MG, McDougle CJ, McCracken JT, Tierney E, Dziura J, Arnold LE, Posey D, Young C, Shah B, Ghuman J, Ritz L, Vitiello B. A prospective open trial of guanfacine in children with pervasive developmental disorders. J Child Adolesc Psychopharmacol. 2006 Oct;16(5):589-98. doi: 10.1089/cap.2006.16.589. PMID 17069547
- [Background] Posey DJ, Wiegand RE, Wilkerson J, Maynard M, Stigler KA, McDougle CJ. Open-label atomoxetine for attention-deficit/ hyperactivity disorder symptoms associated with high-functioning pervasive developmental disorders. J Child Adolesc Psychopharmacol. 2006 Oct;16(5):599-610. doi: 10.1089/cap.2006.16.599. PMID 17069548
- [Background] Kendall AR, Lewy AJ, Sack RL. Effects of aging on the intrinsic circadian period of totally blind humans. J Biol Rhythms. 2001 Feb;16(1):87-95. doi: 10.1177/074873040101600110. PMID 11220783
- [Background] Sack RL, Brandes RW, Kendall AR, Lewy AJ. Entrainment of free-running circadian rhythms by melatonin in blind people. N Engl J Med. 2000 Oct 12;343(15):1070-7. doi: 10.1056/NEJM200010123431503. PMID 11027741
- [Background] Potocki L, Glaze D, Tan DX, Park SS, Kashork CD, Shaffer LG, Reiter RJ, Lupski JR. Circadian rhythm abnormalities of melatonin in Smith-Magenis syndrome. J Med Genet. 2000 Jun;37(6):428-33. doi: 10.1136/jmg.37.6.428. PMID 10851253
- [Background] Pappu AS, Steiner RD, Connor SL, Flavell DP, Lin DS, Hatcher L, Illingworth DR, Connor WE. Feedback inhibition of the cholesterol biosynthetic pathway in patients with Smith-Lemli-Opitz syndrome as demonstrated by urinary mevalonate excretion. J Lipid Res. 2002 Oct;43(10):1661-9. doi: 10.1194/jlr.m200163-jlr200. PMID 12364550